CLINICAL TRIAL: NCT01009463
Title: HZC102871: A 52-week Efficacy and Safety Study to Compare the Effect of Three Dosage Strengths of Fluticasone Furoate/GW642444 Inhalation Powder With GW642444 on the Annual Rate of Exacerbations in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study to Evaluate the Efficacy and Safety of Fluticasone Furoate (FF)/GW642444 Inhalation Powder in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 102871
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2013-08-19 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Safety; FEV1; Efficacy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- FF/GW642444 Inhalation Powder 100/25 mcg QD (Experimental): Inhaled Corticosteroid (ICS)/ Long Acting Beta Agonist(LABA)
  Interventions: Drug: FF/GW642444 Inhalation Powder
- FF/GW642444 Inhalation Powder 200/25 mcg QD (Experimental): Inhaled Corticosteroid (ICS)/ Long Acting Beta Agonist(LABA)
  Interventions: Drug: FF/GW642444 Inhalation Powder
- FF/GW642444 Inhalation Powder 50mcg/25mcg QD (Experimental): Inhaled Corticosteroid (ICS)/ Long Acting Beta Agonist(LABA)
  Interventions: Drug: FF/GW642444 Inhalation Powder
- GW642444 25mcg QD (Experimental): Long Acting Beta Agonist(LABA)
  Interventions: Drug: GW642444 Inhalation Powder

INTERVENTIONS:
Drug: FF/GW642444 Inhalation Powder — Inhaled Corticosteroid (ICS)/ Long Acting Beta Agonist(LABA) delivered within one dry powder inhaler (DPI) device for COPD
  Arms: FF/GW642444 Inhalation Powder 100/25 mcg QD; FF/GW642444 Inhalation Powder 200/25 mcg QD; FF/GW642444 Inhalation Powder 50mcg/25mcg QD
Drug: GW642444 Inhalation Powder — Long Acting Beta Agonist(LABA) Inhalation Powder via DPI
  Arms: GW642444 25mcg QD

SUMMARY:
The Purpose of this study is to assess the efficacy and safety of three strengths of the FF/GW642444 Inhalation Powder in subject with Chronic Obstructive Pulmonary Disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: outpatient
* Informed consent: Subjects must give their signed and dated written informed consent to participate.
* Gender: Male or female subjects A female is eligible to enter and participate in the study if she is of: Non-child bearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g., age appropriate, history of vasomotor symptoms. However in questionable cases, a blood sample with FSH > 40MIU/ml and estradiol <40pg/ml (<140 pmol/L) is confirmatory. OR

Child bearing potential, has a negative pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly (i.e., in accordance with the approved product label and the instructions of the physician for the duration of the study - screening to follow-up contact):

* Complete abstinence from intercourse from screening until the Follow-Up Phone Contact; or
* Male partner is sterile (vasectomy with documentation of azoospermia) prior to female subject entry into the study, and this male partner is the sole partner for that subject; or
* Implants of levonorgestral inserted for at least 1 month prior to the study medication administration but not beyond the third successive year following insertion; or
* Injectable progestogen administered for at least 1 month prior to study medication administration and administered until the Follow-Up Phone Contact; or
* Oral contraceptive (combined or progestogen only) administered for at least one monthly cycle prior to study medication administration; or
* Double barrier method: condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam/gel/film/cream/suppository); or
* An intrauterine device (IUD), inserted by a qualified physician, with published data showing that the highest expected failure rate is less than 1% per year; or
* Estrogenic vaginal ring; or
* Percutaneous contraceptive patches

  * Age: ≥40 years of age at Screening (Visit 1)
  * COPD diagnosis: Subjects with a clinical history of COPD in accordance with the following definition by the American Thoracic Society/European Respiratory Society [Celli, 2004]: COPD is a preventable and treatable disease characterized by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and is associated with an abnormal inflammatory response of the lungs to noxious particles or gases, primarily caused by cigarette smoking. Although COPD affects the lungs, it also produces significant systemic consequences.
  * Tobacco use: Subjects with a current or prior history of ≥10 pack-years of cigarette smoking at Screening (Visit 1). Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. Note: Pipe and/or cigar use cannot be used to calculate pack-year history. Number of pack years = (number of cigarettes per day/20) x number of years smoked
  * Severity of Disease:
* Subject with a measured post-albuterol/salbutamol FEV1/FVC ratio of ≤0.70 at Screening (Visit 1)
* Subjects with a measured post-albuterol/salbutamol FEV1 <70% of predicted normal values calculated (via centralized vendor equipment) using NHANES III reference equations [Hankinson, 1999] at Screening (Visit 1). Post-bronchodilator spirometry will be performed approximately 10-15 minutes after the subject has self-administered 4 inhalations (i.e., total 400mcg) of albuterol/salbutamol via an MDI with a valved-holding chamber. The study provided central spirometry equipment will calculate the FEV1/FVC ratio and FEV1 percent predicted values.

  * History of Exacerbations: A documented history (e.g., medical record verification) of at least one COPD exacerbation in the 12 months prior to Visit 1 that required either oral corticosteroids, antibiotics and/or hospitalization. Prior use of antibiotics alone does not qualify as an exacerbation history unless the use was associated with treatment of worsening symptoms of COPD, such as increased dyspnea, sputum volume, or sputum purulence (color). Subject verbal reports are not acceptable.

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: Subjects with a current diagnosis of asthma. (Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD)
* α1-antitrypsin deficiency: Subjects with α1-antitrypsin deficiency as the underlying cause of COPD
* Other respiratory disorders: Subjects with active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases
* Lung resection: Subjects with lung volume reduction surgery within the 12 months prior to Screening (Visit 1)
* Chest X-ray (or CT scan): Subjects with a chest X-ray (or CT scan) that reveals evidence of clinically significant abnormalities not believed to be due to the presence of COPD. A chest X-ray must be taken at Screening (Visit 1) if a chest X-ray or CT scan is not available within 6 months prior to Visit 1. For sites in Germany, if a chest X-ray (or CT scan) is not available in the 6 months preceding Screening (Visit 1), the subject will not be eligible for the study.
* Risk Factors for Pneumonia: immune suppression (HIV, Lupus, etc) or other risk for pneumonia (e.g. neurological disorders affecting control of the upper airway, such as Parkinson's, Myasthenia Gravis, etc).
* A moderate and severe COPD exacerbation that has not resolved at least 14 days prior to Visit 1 and at least 30 days following the last dose of oral corticosteroids (if applicable).
* Pneumonia and/or moderate and severe COPD exacerbation at Visit 1 Note: Subjects who experience a pneumonia and/or exacerbation at Screening (Visit 1) must be not continue in the study, but may be re-screened at a later time provided the pneumonia and/or COPD exacerbation has resolved prior to the re-screening visit. At the Re-screening Visit, the chest x-ray should confirm resolution of pneumonia. The Re-screening Visit must be conducted at least ≥ 14 days following the resolution date of the exacerbation and/or pneumonia and at least 30 days following the last dose of oral corticosteroids (if applicable).
* Other diseases/abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular (i.e., pacemaker), neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or haematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Peptic Ulcer disease: Subjects with clinically significant peptic ulcer disease that is uncontrolled.
* Hypertension: Subjects with clinically significant hypertension that is uncontrolled.
* Cancer: Subjects with carcinoma that has not been in complete remission for at least 5 years. Carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded if the subject has been considered cured within 5 years since diagnosis.
* Drug/food allergy: Subjects with a history of hypersensitivity to any of the study medications (e.g., beta-agonists, corticosteroid) or components of the inhalation powder (e.g., lactose, magnesium stearate). In addition, subjects with a history of severe milk protein allergy that, in the opinion of the study physician, contraindicates the subject's participation will also be excluded.
* Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years
* Medication prior to spirometry: Subjects who are medically unable to withhold their albuterol/salbutamol and/or their ipratropium for the 4-hour period required prior to spirometry testing at each study visit.
* Additional medication: Unable to stop using certain medications such as bronchodilators and corticosteroids for the protocol-specified times prior to Visit 1 (the Investigator will discuss the specific medications)
* Oxygen therapy: Subjects receiving treatment with long-term oxygen therapy (LTOT) or nocturnal oxygen therapy required for greater than 12 hours a day. Oxygen prn use (i.e., ≤12 hours per day) is not exclusionary.
* Sleep apnea: Subjects with clinically significant sleep apnea who require use of continuous positive airway pressure (CPAP) device or non-invasive positive pressure ventilation (NIPPV) device.
* Pulmonary rehabilitation: Subjects who have participated in the acute phase of a Pulmonary Rehabilitation Program within 4 weeks prior to Screening (Visit 1) or who will enter the acute phase of a Pulmonary Rehabilitation Program during the study. Subjects who are in the maintenance phase of a Pulmonary Rehabilitation Program are not excluded.
* Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* Prior use of study medication/other investigational drugs: Subjects who have previously been randomized to treatment with GW642444 Inhalation Powder in the B2C111045 study, randomized to treatment in the HZC111348 study or have participated in the HZC112207, HZC102871, HZC102970, or HZC110946 studies. Subjects who have received an investigational drug within 30 days of entry into this study (Screening), or within 5 drug half-lives of the investigational drug, whichever is longer.
* Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or immediate family members of the aforementioned are excluded from participating in this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1626 (Actual)
Dates: Start 2009-09-25; Primary Completion 2011-10-01 (Actual); Study Completion 2011-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (166):
- United States (88):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Peoria, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Lincoln, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Palo Alto, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Sepulveda, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Bay Pines, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Austell, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Belleville, Illinois
  - GSK Investigational Site, River Forest, Illinois
  - GSK Investigational Site, Avon, Indiana
  - GSK Investigational Site, Lafayette, Indiana
  - GSK Investigational Site, Muncie, Indiana
  - GSK Investigational Site, Newburgh, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Munfordville, Kentucky
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Saint Joseph, Michigan
  - GSK Investigational Site, Southfield, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Ocean City, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Elizabeth City, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Sellersville, Pennsylvania
  - GSK Investigational Site, Johnston, Rhode Island
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Chester, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenwood, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, New Tazewell, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Boerne, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Kingwood, Texas
  - GSK Investigational Site, Lake Jackson, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Fredericksburg, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Lakewood, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Wenatchee, Washington
- Argentina (3):
  - GSK Investigational Site, Cipolletti, Río Negro Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
- Australia (8):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Cairns, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Daw Park, South Australia
  - GSK Investigational Site, Frankston, Victoria
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (8):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Corunna, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- Chile (3):
  - GSK Investigational Site, Temuco, Región de La Araucania
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Santiago
- Estonia (3):
  - GSK Investigational Site, Rakvere
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (2):
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Italy (9):
  - GSK Investigational Site, Cassano Murge (BA), Apulia
  - GSK Investigational Site, Eboli (SA), Campania
  - GSK Investigational Site, Telese Terme (BN), Campania
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Tradate (VA), Lombardy
  - GSK Investigational Site, Torrette (AN), The Marches
- Mexico (4):
  - GSK Investigational Site, Tijuana, Baja California Norte
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
- Netherlands (12):
  - GSK Investigational Site, Bunnik
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Etten-Leur
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Helmond
  - GSK Investigational Site, Nijverdal
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Sneek
  - GSK Investigational Site, Spijkenisse
  - GSK Investigational Site, Veldhoven
  - GSK Investigational Site, Voerendaal
- Peru (3):
  - GSK Investigational Site, Jesus Maria, Lima region
  - GSK Investigational Site, San Martín de Porres, Lima region
  - GSK Investigational Site, Lima
- Philippines (2):
  - GSK Investigational Site, Dagupan
  - GSK Investigational Site, Quezon City
- South Africa (13):
  - GSK Investigational Site, Cape Town, Gauteng
  - GSK Investigational Site, Mueckelneck, Gauteng
  - GSK Investigational Site, Boksburg North
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Groenkloof
  - GSK Investigational Site, Lynnwood Manor
  - GSK Investigational Site, Lyttleton
  - GSK Investigational Site, Paarl
  - GSK Investigational Site, Panorama
  - GSK Investigational Site, Reiger Park
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Witbank
- Sweden (4):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Höllviken
  - GSK Investigational Site, Kil
  - GSK Investigational Site, Örebro
- United Kingdom (4):
  - GSK Investigational Site, High Heaton, Newcastle Upon Tyne, Tyne & Wear
  - GSK Investigational Site, Doncaster
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Dransfield MT, Bourbeau J, Jones PW, Hanania NA, Mahler DA, Vestbo J, Wachtel A, Martinez FJ, Barnhart F, Sanford L, Lettis S, Crim C, Calverley PM. Once-daily inhaled fluticasone furoate and vilanterol versus vilanterol only for prevention of exacerbations of COPD: two replicate double-blind, parallel-group, randomised controlled trials. Lancet Respir Med. 2013 May;1(3):210-23. doi: 10.1016/S2213-2600(13)70040-7. Epub 2013 Apr 12. PMID 24429127
- [Derived] Largajolli A, Beerahee M, Yang S. Bayesian approach to investigate a two-state mixed model of COPD exacerbations. J Pharmacokinet Pharmacodyn. 2019 Aug;46(4):371-384. doi: 10.1007/s10928-019-09643-6. Epub 2019 Jun 13. PMID 31197640
- [Derived] Hinds DR, DiSantostefano RL, Le HV, Pascoe S. Identification of responders to inhaled corticosteroids in a chronic obstructive pulmonary disease population using cluster analysis. BMJ Open. 2016 Jun 1;6(6):e010099. doi: 10.1136/bmjopen-2015-010099. PMID 27251682
- [Derived] Crim C, Dransfield MT, Bourbeau J, Jones PW, Hanania NA, Mahler DA, Vestbo J, Wachtel A, Martinez FJ, Barnhart F, Lettis S, Calverley PM. Pneumonia risk with inhaled fluticasone furoate and vilanterol compared with vilanterol alone in patients with COPD. Ann Am Thorac Soc. 2015 Jan;12(1):27-34. doi: 10.1513/AnnalsATS.201409-413OC. PMID 25490706
- [Derived] Svedsater H, Dale P, Garrill K, Walker R, Woepse MW. Qualitative assessment of attributes and ease of use of the ELLIPTA dry powder inhaler for delivery of maintenance therapy for asthma and COPD. BMC Pulm Med. 2013 Dec 7;13:72. doi: 10.1186/1471-2466-13-72. PMID 24314123
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 102871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 102871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 102871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 102871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 102871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 102871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 102871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At Visit (V) 1, eligible participants (par.) entered a 4-week, open-label Run-In Period (RIP) to establish a stable Baseline. At V 2, eligible par. were randomized to a 52 week, double-blind Treatment Period. 2631 par. were screened, 2071 par. entered the RIP, and 1626 par. were randomized, out of which 1622 received at >= 1 study treatment dose.
Groups:
- FP/SAL 250/50 µg BID: Participants (Par.) were instructed to take open label Fluticasone Propionate and Salmeterol (FP/SAL) 250/50 microgram (µg) twice daily (BID) from the ACCUHALER/DISKUS, one inhalation each morning and evening with approximately 12 hours between doses. In addition, all par. were provided supplemental albuterol/salbutamol (metered dose inhaler [MDI] and/or nebules) to be used as needed throughout the study.
- VI 25 µg QD: Participants received a Vilanterol (VI) 25 µg dry inhalation powder once daily (QD) in the morning from the Dry Powder Inhaler (DPI) for the duration of the 52 weeks. In addition, all participants were provided supplemental albuterol/salbutamol (MDI and/or nebules) to be used as needed throughout the study.
- FF/VI 50/25 µg QD: Participants received a Fluticasone Furoate/Vilanterol (FF/VI) 50/25 µg inhalation powder QD in the morning from the DPI for the duration of the 52 weeks. In addition, all participants were provided supplemental albuterol/salbutamol (MDI and/or nebules) to be used as needed throughout the study.
- FF/VI 100/25 µg QD: Participants received a FF/VI 100/25 µg inhalation powder QD in the morning from the DPI for the duration of the 52 weeks. In addition, all participants were provided supplemental albuterol/salbutamol (MDI and/or nebules) to be used as needed throughout the study.
- FF/VI 200/25 µg QD: Participants received a FF/VI 200/25 µg inhalation powder QD in the morning from the DPI for the duration of the 52 weeks. In addition, all participants were provided supplemental albuterol/salbutamol (MDI and/or nebules) to be used as needed throughout the study.
Period: 4-week, Open-label Run-In Period
Arm/Group | FP/SAL 250/50 µg BID | VI 25 µg QD | FF/VI 50/25 µg QD | FF/VI 100/25 µg QD | FF/VI 200/25 µg QD
Started | 2071 | 0 | 0 | 0 | 0
Completed | 1622 | 0 | 0 | 0 | 0
Not Completed | 449 | 0 | 0 | 0 | 0
Not completed — Did Not Meet Continuation Criteria | 373 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 10 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 6 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 10 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 50 | 0 | 0 | 0 | 0
Period: 52-week, Double-blind Treatment Period
Arm/Group | FP/SAL 250/50 µg BID | VI 25 µg QD | FF/VI 50/25 µg QD | FF/VI 100/25 µg QD | FF/VI 200/25 µg QD
Started | 0 | 409 | 408 | 403 | 402
Completed the Treatment Period | 0 | 295 (Par. completed the treatment period if they attended the last treatment visit (Visit 11).) | 318 (Par. completed the treatment period if they attended the last treatment visit (Visit 11).) | 314 (Par. completed the treatment period if they attended the last treatment visit (Visit 11).) | 303 (Par. completed the treatment period if they attended the last treatment visit (Visit 11).)
Completed | 0 | 294 (Par. completed the study if they completed the treatment period and safety follow-up phone contact.) | 315 (Par. completed the study if they completed the treatment period and safety follow-up phone contact.) | 312 (Par. completed the study if they completed the treatment period and safety follow-up phone contact.) | 301 (Par. completed the study if they completed the treatment period and safety follow-up phone contact.)
Not Completed | 0 | 115 | 93 | 91 | 101
Not completed — Adverse Event | 0 | 22 | 25 | 29 | 31
Not completed — Withdrawal by Subject | 0 | 34 | 18 | 17 | 22
Not completed — Lack of Efficacy | 0 | 24 | 16 | 11 | 18
Not completed — Protocol Violation | 0 | 8 | 7 | 8 | 7
Not completed — Met Protocol-Defined Stopping Criteria | 0 | 10 | 14 | 13 | 10
Not completed — Study Closed/Terminated | 0 | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 11 | 7 | 6 | 5
Not completed — Physician Decision | 0 | 4 | 6 | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VI 25 µg QD | FF/VI 50/25 µg QD | FF/VI 100/25 µg QD | FF/VI 200/25 µg QD | Total
Number analyzed (Participants) | 409 | 408 | 403 | 402 | 1622
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (9.43) | 63.6 (9.06) | 63.6 (9.06) | 63.8 (9.30) | 63.6 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170 | 163 | 172 | 153 | 658
  Male | 239 | 245 | 231 | 249 | 964
Race/Ethnicity, Customized [Number; unit: participants]
  White | 331 | 334 | 332 | 324 | 1321
  African American/ African Heritage | 9 | 8 | 6 | 9 | 32
  Asian | 39 | 37 | 37 | 41 | 154
  American Indian or Alaska Native & White | 19 | 16 | 19 | 15 | 69
  Asian & White | 0 | 1 | 0 | 0 | 1
  American Indian or Alaska Native | 10 | 12 | 9 | 12 | 43
  Unknown | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Moderate and Severe COPD Exacerbations Expressed as Least Square Mean
Description: The annual rate of moderate and severe chronic obstructive pulmonary disease (COPD) exacerbations during the treatment (trt) period (per participant [par.] per year) was assessed. An exacerbation of COPD, is defined as the worsening of two or more major symptoms (dyspnea, sputum volume, sputum purulence [color]) for at least two consecutive days; or the worsening of any one major symptom together with any one of the minor symptoms (sore throat, cold, fever without other cause, increased cough, increased wheeze) for at least two consecutive days. The COPD exacerbation was categorized as mild, moderate and severe by the investigator. Mild: worsening symptoms of COPD that were self-managed by the par. without the use of oral corticosteroids or antibiotics; Moderate: worsening symptoms of COPD that required treatment with oral corticosteroids and/or antibiotics; Severe: worsening symptoms of COPD that required treatment with in-patient hospitalization.
Time Frame: From the start of the double blinded study medication until Visit 11 (Week 52)/Early Withdrawal
Population: Intent-to-Treat (ITT) Population: all par. randomized who received at least 1 dose of study drug and with available data for analysis. Analysis used a negative binomial regression model with covariates of trt, smoking status at Screening, Baseline pre-dose Day 1 % predicted FEV1 and region and with logarithm of time on trt as an offset variable.
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations per participant per year
Arm/Group | VI 25 µg QD | FF/VI 50/25 µg QD | FF/VI 100/25 µg QD | FF/VI 200/25 µg QD
Number analyzed (Participants) | 409 | 408 | 403 | 402
Exacerbations per participant per year | 1.05 [0.92 to 1.21] | 0.92 [0.80 to 1.06] | 0.70 [0.60 to 0.81] | 0.90 [0.78 to 1.04]
Statistical Analysis 1: Comparison: VI 25 µg QD vs FF/VI 50/25 µg QD; Test type: Superiority or Other; p = 0.181, Generalized Linear Model; Assuming Negative Binomial distribution with logarithm of time on treatment as an offset variable; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.72 to 1.06]
Statistical Analysis 2: Comparison: VI 25 µg QD vs FF/VI 100/25 µg QD; Test type: Superiority or Other; p < 0.001, Generalized Linear Model — Nominal p-value; Assuming Negative Binomial distribution with logarithm of time on treatment as an offset variable; Risk Ratio (RR) = 0.66, 95% CI 2-sided [0.54 to 0.81]
Statistical Analysis 3: Comparison: VI 25 µg QD vs FF/VI 200/25 µg QD; Test type: Superiority or Other; p = 0.109, Generalized Linear Model; Assuming Negative Binomial distribution with logarithm of time on treatment as an offset variable; Risk Ratio (RR) = 0.85, 95% CI 2-sided [0.70 to 1.04]

2. Secondary Outcome: Time to First Occurrence of Moderate or Severe COPD Exacerbation
Description: Time to first occurrence analyzed by using a Cox proportional hazards model with covariates of treatment, smoking status at screening (stratum), baseline disease severity (pre-dose Day 1 % predicted FEV1) and centre grouping. An exacerbation of COPD is defined as the worsening of two or more major symptoms (dyspnea, sputum volume, sputum purulence [color]) for at least two consecutive days; or the worsening of any one major symptom together with any one of the minor symptoms (sore throat, cold, fever without other cause, increased cough, increased wheeze) for at least two consecutive days. A moderate exacerbation is defined as worsening symptoms of COPD that required treatment with oral corticosteroids and/or antibiotics. A severe exacerbation is defined as worsening symptoms of COPD that required treatment with in-patient hospitalization. The number of participants with a moderate or severe COPD exacerbation while on treatment are presented.
Time Frame: From the start of the double blind study medication until Visit 11 (Week 52)/Early Withdrawal
Population: ITT Population
Measure: Number; unit: Participants
Groups:
- VI 25 µg QD: Participants received a Vilanterol (VI) 25 µg dry inhalation powder once daily (QD) in the morning from the Dry Powder Inhaler (DPI) for the duration of the 52 weeks. In addition, all participants were provided supplemental albuterol/salbutamol (MDI and/or nebules) to be used as needed throughout the study. )
Arm/Group | VI 25 µg QD | FF/VI 50/25 µg QD | FF/VI 100/25 µg QD | FF/VI 200/25 µg QD
Number analyzed (Participants) | 409 | 408 | 403 | 402
Participants | 202 | 190 | 160 | 178
Statistical Analysis 1: Comparison: VI 25 µg QD vs FF/VI 50/25 µg QD; Test type: Superiority or Other; p = 0.430, Regression, Cox; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.76 to 1.13]
Statistical Analysis 2: Comparison: VI 25 µg QD vs FF/VI 100/25 µg QD; Test type: Superiority or Other; p = 0.002, Regression, Cox — Nominal p-value; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.59 to 0.89]
Statistical Analysis 3: Comparison: VI 25 µg QD vs FF/VI 200/25 µg QD; Test type: Superiority or Other; p = 0.114, Regression, Cox; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.69 to 1.04]

3. Secondary Outcome: Annual Rate of Exacerbations Requiring Systemic/Oral Corticosteroids Expressed as Least Square Mean
Description: The annual rate of COPD exacerbations during the treatment period (per participant per year) that required systemic/oral corticosteroids was assessed. An exacerbation of COPD is defined as the worsening of two or more major symptoms (dyspnea, sputum volume, sputum purulence [color]) for at least two consecutive days; or the worsening of any one major symptom together with any one of the minor symptom (sore throat, cold, fever without other cause, increased cough, increased wheeze) for at least two consecutive days. The COPD exacerbation was categorized as mild, moderate, and severe by the investigator. Mild: worsening symptoms of COPD that were self-managed by the participant. Mild exacerbations were not associated with the use of oral corticosteroids or antibiotics. Moderate: worsening symptoms of COPD that required treatment with oral corticosteroids and/or antibiotics. Severe: worsening symptoms of COPD that required treatment with in-patient hospitalization.
Time Frame: From the start of the double blind study medication until Visit 11 (Week 52)/Early Withdrawal
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations per participant per year
Arm/Group | VI 25 µg QD | FF/VI 50/25 µg QD | FF/VI 100/25 µg QD | FF/VI 200/25 µg QD
Number analyzed (Participants) | 409 | 408 | 403 | 402
Exacerbations per participant per year | 0.84 [0.72 to 0.98] | 0.71 [0.60 to 0.83] | 0.52 [0.44 to 0.62] | 0.68 [0.57 to 0.80]
Statistical Analysis 1: Comparison: VI 25 µg QD vs FF/VI 50/25 µg QD; Test type: Superiority or Other; p = 0.125, Generalized Linear Model; Assuming Negative Binomial distribution with logarithm of time on treatment as an offset variable; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.67 to 1.05]
Statistical Analysis 2: Comparison: VI 25 µg QD vs FF/VI 100/25 µg QD; Test type: Superiority or Other; p < 0.001, Generalized Linear Model — Nominal p-value; Assuming Negative Binomial distribution with logarithm of time on treatment as an offset variable; Risk Ratio (RR) = 0.62, 95% CI 2-sided [0.49 to 0.78]
Statistical Analysis 3: Comparison: VI 25 µg QD vs FF/VI 200/25 µg QD; Test type: Superiority or Other; p = 0.064, Generalized Linear Model; Assuming Negative Binomial distribution with logarithm of time on treatment as an offset variable; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.64 to 1.01]

4. Secondary Outcome: Change From Baseline in Trough FEV1 at Week 52 (Visit 11)
Description: Pulmonary function was measured by forced expiratory volume in one second (FEV1). Trough FEV1 was defined as the 24-hour post-dose FEV1 assessment, which was obtained at each visit. Analysis performed using a repeated measures model with covariates of treatment, smoking status at Screening (stratum), baseline (pre-dose Day 1), centre grouping, Week, Week by Baseline, and Week by treatment interactions.
Time Frame: Baseline to Visit 11 (Week 52)/Early Withdrawal
Population: ITT Population. Number of participants presented represent those with data available at the time point being presented, however all participants in the ITT population without missing covariate information and with at least one post Baseline measurement are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | VI 25 µg QD | FF/VI 50/25 µg QD | FF/VI 100/25 µg QD | FF/VI 200/25 µg QD
Number analyzed (Participants) | 291 | 308 | 310 | 289
Liters | -0.040 (0.0114) | 0.000 (0.0112) | 0.018 (0.0112) | 0.024 (0.0114)
Statistical Analysis 1: Comparison: VI 25 µg QD vs FF/VI 50/25 µg QD; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.041, 95% CI 2-sided [0.009 to 0.072]
Statistical Analysis 2: Comparison: VI 25 µg QD vs FF/VI 100/25 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.058, 95% CI 2-sided [0.027 to 0.090]
Statistical Analysis 3: Comparison: VI 25 µg QD vs FF/VI 200/25 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.064, 95% CI 2-sided [0.033 to 0.096]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs will be collected from Baseline to the end of the treatment period (up to 52 weeks).
Description: SAEs and non-serious adverse events are reported for members of the Intent-to-Treat Population, comprised of all randomized participants who received at least one dose of study medication during the treatment period.
Arm/Group | VI 25 µg QD | FF/VI 50/25 µg QD | FF/VI 100/25 µg QD | FF/VI 200/25 µg QD
Serious Adverse Events (participants affected / at risk) | 60/409 | 65/408 | 56/403 | 63/402
Other Adverse Events (participants affected / at risk) | 197/409 | 227/408 | 221/403 | 225/402
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VI 25 µg QD (N=409) | FF/VI 50/25 µg QD (N=408) | FF/VI 100/25 µg QD (N=403) | FF/VI 200/25 µg QD (N=402)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 28 | 27 | 26 | 30
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 12 | 9 | 12
Cellulitis (Infections and infestations) | 2 | 0 | 4 | 0
Infective exacerbation of chronic obstructive airway disease (Infections and infestations) | 2 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Bone tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
H1N1 influenza (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 0 | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 2 | 2 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 2 | 0 | 0
Angina unstable (Cardiac disorders) | 2 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery thrombosis (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0
AE Term: Salivary gland enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant hepatobiliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 2 | 3
Syncope (Nervous system disorders) | 2 | 1 | 0 | 0
Carotid artery aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0
Shock (Vascular disorders) | 1 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 2 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 3 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VI 25 µg QD (N=409) | FF/VI 50/25 µg QD (N=408) | FF/VI 100/25 µg QD (N=403) | FF/VI 200/25 µg QD (N=402)
Nasopharyngitis (Infections and infestations) | 54 | 58 | 60 | 76
Upper respiratory tract infection (Infections and infestations) | 45 | 47 | 51 | 39
Oral candidiasis (Infections and infestations) | 21 | 39 | 34 | 36
Bronchitis (Infections and infestations) | 20 | 13 | 21 | 23
Sinusitis (Infections and infestations) | 17 | 21 | 22 | 13
Pneumonia (Infections and infestations) | 10 | 17 | 16 | 16
Influenza (Infections and infestations) | 21 | 10 | 13 | 13
Pharyngitis (Infections and infestations) | 14 | 8 | 14 | 16
Urinary tract infection (Infections and infestations) | 7 | 16 | 10 | 17
Rhinitis (Infections and infestations) | 6 | 9 | 10 | 15
Oropharyngeal candidiasis (Infections and infestations) | 2 | 14 | 7 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 21 | 24 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 13 | 16 | 13
Headache (Nervous system disorders) | 30 | 27 | 25 | 34
Dizziness (Nervous system disorders) | 8 | 13 | 5 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 21 | 16 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 7 | 14 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 13 | 6 | 4
Diarrhoea (Gastrointestinal disorders) | 15 | 12 | 8 | 15
Nausea (Gastrointestinal disorders) | 10 | 24 | 7 | 10
Hypertension (Vascular disorders) | 6 | 15 | 19 | 12
Pyrexia (General disorders) | 5 | 17 | 10 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.